CLINICAL TRIAL: NCT03669549
Title: A Multicenter Dose-Titration Open-Label Study of Nevanimibe Hydrochloride for the Treatment of Classic Congenital Adrenal Hyperplasia
Brief Title: Nevanimibe HCl for the Treatment of Classic CAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following an interim data review, further investment in nevanimibe has been discontinued
Sponsor: Millendo Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Organization: Millendo Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATR-101-202
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: CAH; nevanimibe
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nevanimibe hydrochloride (Experimental): Ascending dose level of oral nevanimibe hydrochloride beginning with 500 mg BID up to 2000 mg BID
  Interventions: Drug: Nevanimibe hydrochloride

INTERVENTIONS:
Drug: Nevanimibe hydrochloride — During the 16-week treatment period, all subjects will begin dosing with nevanimibe HCl 500 mg BID and be dose titrated to 1000 mg BID, 1500 mg BID, and 2000 mg BID as needed based on serum 17-OHP assessments every 4 weeks.

SUMMARY:
This is a multicenter, intra-subject dose-titration open-label study of nevanimibe hydrochloride (HCl) for the treatment of classic congenital adrenal hyperplasia (CAH). Following a Screening Period of approximately 2-14 weeks, eligible subjects will enter a Baseline Period of approximately 2-8 weeks and then a 16-week Treatment Period. It is anticipated that the overall duration of the study per subject will range from 24-42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented historical diagnosis of classic CAH due to 21-hydroxylase deficiency and/or historical documentation of elevated 17-OHP
* Chronic glucocorticoid replacement therapy for at least 6 consecutive months prior to screening
* Stable glucocorticoid and mineralocorticoid regimen for at least 4 weeks prior to screening and throughout the treatment period of the study

Exclusion Criteria:

* Nonclassic CAH
* Other causes of adrenal insufficiency
* HIV, hepatitis B, or hepatitis C
* AST or ALT >2x ULN, bilirubin or serum creatinine >1.5x ULN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Brazil (3):
  - University of Ribeirão Preto, Medicine Faculty (Faculdade de Medicina) of Ribeirão Preto, Ribeirão Preto
  - Universidade Federal de São Paulo, Escola Paulista de Medicina, São Paulo
  - Hospital das Clínicas da FMUSP - Prédio do Instituto Central, São Paulo
- Institute of Endocrinology, Prague, Czechia
- Hospital Pitié-Salpetrière, Paris, France
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Beilinson Hospital, Petah Tikva
  - Tel-Aviv-Sourasky Medical Center, Tel Aviv
- Spain (3):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - University Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White PC. Emerging treatment for congenital adrenal hyperplasia. Curr Opin Endocrinol Diabetes Obes. 2022 Jun 1;29(3):271-276. doi: 10.1097/MED.0000000000000723. PMID 35283460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global Amendment 1:
  Approximately 20-24 adults with a documented history of classic CAH will be enrolled
  Global Amendment 2:
  Approximately 20-24 evaluable adults with a documented history of classic CAH will be enrolled 20-24 patients planned, 15 patients analyzed
Pre-assignment Details: Screening Period of 2-14 weeks After signing informed consent, patients with classic CAH entered the Screening Period to assess preliminary eligibility for the study based on the inclusion and exclusion criteria. In addition, pertinent information was collected such as past medical history, demographic data, and prior and current medications.
Groups:
- Nevanimibe HCl: Ascending dose level of oral nevanimibe hydrochloride beginning with 500 mg BID up to 2000 mg BID
  Nevanimibe hydrochloride: During the 16-week treatment period, all subjects will begin dosing with nevanimibe HCl 500 mg BID and be dose titrated to 1000 mg BID, 1500 mg BID, and 2000 mg BID as needed based on serum 17-OHP assessments every 4 weeks.
Period: Overall Study
Arm/Group | Nevanimibe HCl
Started | 15
Completed | 9
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Study terminated by the Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nevanimibe HCl
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 2
  Brazil | 1
  Israel | 4
  France | 2
  Spain | 6
Baseline serum 17-hydroxyprogesterone [Mean (Standard Deviation); unit: ng/dL] | 10644.1 (10618.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Serum 17-OHP Targets
Description: The primary efficacy endpoint was the overall response rate within each cohort, defined as the percentage of patients achieving serum 17-OHP targets as follows:
  * Men and postmenopausal women: 17-OHP ≤ 2x ULN
  * Premenopausal women:
    * Follicular phase: 17-OHP ≤ 2x follicular phase ULN
    * Luteal phase: 17-OHP ≤ (2x follicular phase ULN + (luteal phase ULN - follicular phase ULN))
Time Frame: Through Day 113
Measure: Number; unit: percent
Arm/Group | Nevanimibe HCl
Number analyzed (Participants) | 15
percent | 7.1

ADVERSE EVENTS:
Time Frame: From the time of informed consent through treatment period and until 30 days after the last dose of study drug
Groups:
- Nevanimibe HCl Dose Level: <500 mg BID; Nevanimibe HCl Dose Level:500 to <1000 mg BID; Nevanimibe HCl Dose Level: 1000 to <1500 mg BID; Nevanimibe HCl Dose Level: 1500 to <2000 mg BID; Nevanimibe HCl Dose Level:2000 mg BID: Ascending dose level of oral nevanimibe hydrochloride beginning with 500 mg BID up to 2000 mg BID
  Nevanimibe hydrochloride: During the 16-week treatment period, all subjects will begin dosing with nevanimibe HCl 500 mg BID and be dose titrated to 1000 mg BID, 1500 mg BID, and 2000 mg BID as needed based on serum 17-OHP assessments every 4 weeks.
Arm/Group | Nevanimibe HCl Dose Level: <500 mg BID | Nevanimibe HCl Dose Level:500 to <1000 mg BID | Nevanimibe HCl Dose Level: 1000 to <1500 mg BID | Nevanimibe HCl Dose Level: 1500 to <2000 mg BID | Nevanimibe HCl Dose Level:2000 mg BID
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/5 | 0/14 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/5 | 1/14 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/14 | 5/5 | 8/14 | 7/9 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nevanimibe HCl Dose Level: <500 mg BID (N=14) | Nevanimibe HCl Dose Level:500 to <1000 mg BID (N=5) | Nevanimibe HCl Dose Level: 1000 to <1500 mg BID (N=14) | Nevanimibe HCl Dose Level: 1500 to <2000 mg BID (N=9) | Nevanimibe HCl Dose Level:2000 mg BID (N=9)
Uroinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nevanimibe HCl Dose Level: <500 mg BID (N=14) | Nevanimibe HCl Dose Level:500 to <1000 mg BID (N=5) | Nevanimibe HCl Dose Level: 1000 to <1500 mg BID (N=14) | Nevanimibe HCl Dose Level: 1500 to <2000 mg BID (N=9) | Nevanimibe HCl Dose Level:2000 mg BID (N=9)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia, Chest pain, Fatigue, Noncardiac chest pain, Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Insomnia, Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough, Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention, Headache, Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort, Diarrhoea, Dyspepsia, Flatulence, Gingival bleeding, Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Dysuria, Hypertonic bladder, Micturition urgency, Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Acne, Eczema, Pruritus, Rash, Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis, Nasopharyngitis, Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Nevanimibe hydrochloride administered orally at doses of 500-2000 mg BID for up to 16 weeks in the first 10 evaluable patients did not result in sufficient efficacy. The Sponsor has decided to refrain from further development at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT03669549/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03669549/SAP_001.pdf